CLINICAL TRIAL: NCT06167395
Title: Randomized Clinical Trial to Analyze the Efficacy of Chronic Intake of Different Doses of a β-alanine Supplement on Aerobic Performance in Recreational Long-Distance Road Cyclists
Brief Title: Study to Analyze the Aerobic Performance Efficacy of Chronic Intake With a β-alanine Supplement in Recreational Cyclists
Acronym: B-AC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCAMCFE-00031
Record Dates: First submitted 2023-12-02; First posted 2023-12-12 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-11

CONDITIONS: Beta Alanine Supplementation
Keywords: Aerobic Performance; Beta Alanine; Supplementation
MeSH Terms: interventions — beta-Alanine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beta Alanine high dose (Experimental): Consumption for 30 days.
  Interventions: Dietary Supplement: Beta Alanine high dose
- Beta Alanine low dose (Experimental): Consumption for 30 days.
  Interventions: Dietary Supplement: Beta Alanine low dose
- Control group (Placebo Comparator): Consumption for 30 days.
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Beta Alanine high dose — Subjects should consume 4 intakes of 5 g of beta alanine every 3 hours each day.
  Arms: Beta Alanine high dose
Dietary Supplement: Beta Alanine low dose — Subjects should consume 4 intakes of 2,5 g of beta alanine every 3 hours each day.
  Arms: Beta Alanine low dose
Dietary Supplement: Control product — Subjects should consume 4 intakes of 2,5 g of wheat semolina every 3 hours each day.
  Arms: Control group

SUMMARY:
Randomized, controlled, double-blind, double-blind clinical trial, with three parallel arms depending on the product consumed (experimental product dose 1 and dose 2 and placebo product) and single-center, to measure the efficacy of a sustained release beta alanine on the aerobic performance efficacy in recreational cyclist

DETAILED DESCRIPTION:
Subjects meeting the selection criteria will be randomly assigned to each of the study groups (investigational product dose 1 or dose 2, or placebo, depending on the group to which they have been assigned).

The product to be consumed is beta alanine. Participants will consume the product for 30 days. They will have to take 4 intakes every three hours, being the first intake two hours after waking up.

The study subjects will have to make 2 visits to the laboratory. At the first and last visit, their aerobic performance will be evaluated by an incremental test to exhaustion with gas analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male cyclists with more than two years of cycling experience.
* Perform tests without fatigue.
* Road bike training at least twice a week.

Exclusion Criteria:

* Participants with chronic illness.
* Have a long-term injury that prevents you from training in the previous month.
* Inability to understand informed consent.
* Have consumed beta alanine in the three years prior to the start of the study.
* Consumption of other supplements that may alter performance.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Power | Change in performance after 30 days of product consumption
  Measured using a cyclus 2 roller.
Distance | Change in performance after 30 days of product consumption
  Measured using a cyclus 2 roller.

SECONDARY OUTCOMES:
Anaerobic treshold | It will be measured twice, once at baseline or at the end of the study after 30 days.
  Through a stress test with gas analysis
Maximum oxygen consumption | It will be measured twice, once at baseline or at the end of the study after 30 days.
  Through a stress test with gas analysis
Aerobic threshold | It will be measured twice, once at baseline or at the end of the study after 30 days.
  Through a stress test with gas analysis
Microcapillary blood | It will be measured twice, once at baseline or at the end of the study after 30 days.
  This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood.
Lactate | It will be measured twice, once at baseline or at the end of the study after 30 days.
  Lactate levels will be measured using the Lactate Pro 2
Heart Rate | It will be measured twice, once at baseline or at the end of the study after 30 days.
  The heart rate will be evaluated by means of a heart rate strap.
Fatigue | It will be measured twice, once at baseline or at the end of the study after 30 days.
  Rate of perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain